CLINICAL TRIAL: NCT04757103
Title: Surgical Approach for Retro-rectal Tumors: a Retrospective Bicentric Cohort (SART Cohort)
Brief Title: Surgical Approach for Retrorectal Tumors Cohort
Acronym: SART cohort
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0093
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Malignant Tumor
Keywords: Retrorectal tumor; Tail gut cyst; Benign tumor; Mini-invasive approach; Open approach; Perineal approach
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Above S3: Lesion located above the third sacral vertebra
  Interventions: Procedure: Resection of the retrorectal tumor
- Below S3: Lesion located below the third sacral vertebra
  Interventions: Procedure: Resection of the retrorectal tumor

INTERVENTIONS:
Procedure: Resection of the retrorectal tumor — Surgical resection of the retrorectal mass

SUMMARY:
Aim of the study :

To evaluate postoperative outcomes of all surgical approach for retrorectal tumors.

Methods :

From 2005 to 2020, all consecutive patients who underwent surgery for a retrorectal tumor in two referral tertiary center were prospectively collected.

Considering our exlusion criterias, data from XX patients were analyzed. The cohort was separated into 2 groups according to tumor localization regarding the third sacral vertebra.

Short and longterm outcomes were compared between the two groups.

Primary outcome :

90 days postoperative morbidity rate

DETAILED DESCRIPTION:
Retro-rectal tumors are a group of heterogeneous and rare lesions. The actual incidence has been estimated to be approximately one case per 40,000 admissions. It is most often a benign tumor that affects young women and the origin is congenital in 60% of cases. The most common benign lesion is a tailgut cyst. Chordoma is the most common malignant lesion. They are mostly asymptomatic or pauci-symptomatic. This is why their diagnosis is regularly accidentaly after a morphological examination such as an abdominal ultrasound or a CT scan. MRI is the gold standard for determining the structure of the lesion, its origin, its topography, its extension in relation to adjacent organs, parameters that are essential to define the type of surgery and its approach.

When a retro-rectal tumor is diagnosed, the standard treatment is surgical resection. A biopsy is not helpful if there is no suspicion of a degenerate lesion. Usually, lesions located under the third sacral vertebra (S3) are approached by dorsal transsacrococcygeal, perineal or combined approach (abdominal and perineal approach) while those located above S3 the approach is abdominal (laparotomy or laparoscopy). As these lesions are, in the majority of cases, benign, the functional impact of surgery is essential. Based on our experience in minimally invasive surgery and in particular in retro-rectal tumors, laparoscopy has become our first-line approach regardless of the location of the lesion compared to S3. Our hypothesis is that the minimally invasive approach is reliable, safe and allows satisfactory histological results to be obtained while limiting postoperative pain and functional sequelae.

ELIGIBILITY:
Inclusion criteria:

* Patient presenting a retrorectal tumor
* Surgical procedure between 01/01/2005 and 31/12/2020

Exclusion criteria:

* age < 18 years old
* Patients presenting a rectal tumor
* Patients presenting a rectal duplication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a retrorectal tumor who underwent surgical excision
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity rate | 90 days
  Postoperative morbidity according to Clavien Dindo

SECONDARY OUTCOMES:
Mortality rate | 90 days
  Mortality rate
Reoperation rate | 90 days
  Any reoperation linked to surgical resection of the retrorectal tumor
Quality of surgical resection | 90 days
  Evaluation of surgical margins according to pathological examination
Conversion to open approach | 90 days
  Conversion to laparotomy in case of mini-invasive approach
Rate of functional outcomes | 90 days
  Evaluation of fecal
Rate of functional outcomes | 90 days
  Evaluation urinary functions
Functional outcomes | 90 days
  Evaluation of sexual functions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bardol, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC